CLINICAL TRIAL: NCT05728398
Title: Music in Interventional Radiology Procedures: Effect on Patient and Staff Experience
Brief Title: Music in Interventional Radiology Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WESTERNU_IR 001
Record Dates: First submitted 2022-07-12; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Patient Satisfaction
Keywords: Interventional radiology; Music; procedure sedation; patient experience
MeSH Terms: conditions — Patient Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention Group (Active Comparator): Participants randomized to receive music intervention during interventional radiology procedure.
  Interventions: Other: Music
- No Music Comparator Group (Sham Comparator): Participants randomized to have no music played during interventional radiology procedure.
  Interventions: Other: No Music

INTERVENTIONS:
Other: Music — Music played within the fluoroscopy suite during an interventional radiology procedure.
  Arms: Music Intervention Group
Other: No Music — No music played within the fluoroscopy suite during an interventional radiology procedure.
  Arms: No Music Comparator Group

SUMMARY:
The use of music as medical therapy for the treatment of mental health conditions like depression and anxiety is well established. Furthermore, music is sometimes played in operating rooms and several small single center studies done during cardiology and interventional radiology procedures have demonstrated that the use of music can decrease in the use of sedation medications, pain, and anxiety during the procedures.

These past studies have only looked at the impact on the participants, as the music was delivered to the participants only through headphones. This means that the impact of music on the healthcare team was not studied. However, separate systematic literature reviews on the impact of playing music in operating rooms during surgical procedures have highlighted some positive effects music has on the surgeon and the surgical team.

The purpose of this study is to evaluate the effects of playing music during interventional radiology procedures on the participants and the healthcare team. One way of studying this is to compare the responses and experience of participants and healthcare team that hear ambient music during the procedure with those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an out-patient or non-emergent in-patient interventional radiology procedure

Exclusion Criteria:

* Participants unable to consent or complete survey information
* Participants receiving procedures under general anesthesia
* Participants unable to receive IV conscious sedation
* Emergent cases or those performed outside of routine hospital hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Procedural Sedation required | Intra-procedure
  Dosage of Fentanyl and Midazolam required during interventional radiology procedure

SECONDARY OUTCOMES:
Participant intra-procedural anxiety | Intra-procedure
  Assess peri-procedural anxiety using State-Trait Anxiety Inventory scale
Participant procedural pain | Immediately post-procedure
  Participant qualitative assessment of procedural pain using Visual Analog Scale (VAS)
Participant Procedural Experience | Immediately post-procedure
  Participant Experience qualitative assessment using Likert scale
Interventional radiology procedure length | Intra-procedure
  Measure the total time required to perform the IR procedure
Healthcare team experience | Immediately post-procedure
  Assess procedural healthcare team's (physician, IR nurse, & IR technologist) perceived impact of music on the procedure experience (Likert scale)